CLINICAL TRIAL: NCT06812481
Title: Anticholinergic Drug Use in Patients With Rheumatoid Arthritis and Its Effects on Fracture Risk
Brief Title: Anticholinergic Burden and Osteoporosis in Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Bilal Uysal, Assistant professor, Balikesir University
Other Study IDs: RA anticholinergic load
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis (RA); Anticholinergic Adverse Reaction; Fractures, Bone
Keywords: Rheumatoid arthritis; anticholinergic load; risk of fracture
MeSH Terms: conditions — Arthritis, Rheumatoid; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: ACB risk score of 3 or more (high risk).
  Interventions: Other: Anticholinergic load was calculated using anticholinergic cognitive load (ACB)
- group 2: ACB risk score of less than 3 (low risk)
  Interventions: Other: Anticholinergic load was calculated using anticholinergic cognitive load (ACB)

INTERVENTIONS:
Other: Anticholinergic load was calculated using anticholinergic cognitive load (ACB) — Bone mineral density was measured using a Dual Energy X-ray Absorptiometry (DEXA) device.
  Fracture Risk Assessed with Fracture Risk Assessment Tool (FRAX).

SUMMARY:
Background: Rheumatoid arthritis (RA) is a chronic, progressive, inflammatory rheumatological disease. Use of corticosteroids for more than 3 months in RA treatment is considered an important risk factor in terms of developing secondary osteoporosis and increasing the risk of fracture. The cumulative effect of taking one or more drugs with anticholinergic properties is called anticholinergic load. It is stated that anticholinergic load also increases the risk of fracture in individuals. The aim of this study is to investigate the effects of drugs used by patients with Rheumatoid Arthritis (RA) on anticholinergic load and fracture risk. The Fracture Risk Assessment Tool (FRAX) will be used to assess fracture risk in patients.

Materials and methods: The study was planned as a prospective cohort study. The study will included 100 patients who were followed up as outpatients with rheumatoid arthritis diagnosis in the physical medicine and rehabilitation clinic between 2024-2025. Patients of both genders and over 18 years of age diagnosed with rheumatoid arthritis will be included in the study. Patients with systemic diseases or medications affecting bone metabolism and those with metallic materials in the hip or lumbar vertebrae affecting bone mineral density measurement will be excluded from the study. Demographic characteristics, systemic diseases, medications used, bone density measurement and blood test values of the patients will be recorded.

Patients taking multiple medications with anticholinergic effects create an anticholinergic burden. The Anticholinergic Drug Scale, Anticholinergic Cognitive Burden Scale and Anticholinergic Risk Scale will be used to measure anticholinergic burden in the study.

DETAILED DESCRIPTION:
It will be conducted in Balıkesir University, Faculty of Medicine, Health Practice and Research Hospital, Department of Physical Medicine and Rehabilitation.

The study planned to include patients with rheumatoid arthritis classified according to the 2010 American College of Rheumatology/European League Against Rheumatology (ACR/EULAR) criteria. The study will be conducted on patients diagnosed with rheumatoid arthritis and followed up in physical medicine and rehabilitation outpatient clinics.

Bone mineral density measurement (DEXA), urea, creatinine, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, calcium, phosphorus, thyroid stimulating hormone, free thyroxine, parathyroid hormone and 25-OH vitamin D levels in routine examinations of the patients within the last year and the medications used will be obtained from the patient files and recorded.

Patients taking multiple medications with anticholinergic effects create an anticholinergic burden. Several tools have been developed to estimate the cumulative effects of drugs with anticholinergic effects in individuals. They are based on either expert consensus, serum anticholinergic activity or pharmacological principles. The Anticholinergic Drug Scale, Anticholinergic Cognitive Burden Scale and Anticholinergic Risk Scale, which are widely used to measure anticholinergic burden, will be used in the study.

The Fracture Risk Assessment Tool (FRAX) will be used to assess fracture risk in patients. The University of Sheffield launched the FRAX tool in 2008 (Center for Metabolic Bone Diseases, University of Sheffield, UK).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis

Exclusion Criteria:

* Kemik metabolizmasını etkileyen sistemik hastalıkları veya ilaçları kullanan hastalar,
* Kemik mineral yoğunluk ölçümünü etkileyen kalça veya lomber vertebralarda metalik materyalleri olan hastalar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Anticholinergic Cognitive Load (ACB) | 1 week after the start of the study
  The ACB score is a score that determines the impact of anticholinergic medications. ACB is a scale that was introduced in 2008 and is widely used to estimate anticholinergic burden and its relationship with cognitive impairment. ACB is the most easily accessible and most frequently used scale in practice. The scale scores between 0 and 3 according to the affinity of the drugs to muscarinic receptors and their effects on cognition. 0 is no burden; a score of 3 or above is considered high risk. The anticholinergic burden of 88 drugs is calculated in the ACB score.
The Anticholinergic Risk Scale (ARS) | 1 week after the start of the study
  The Anticholinergic Risk Scale (ARS) is used to estimate the extent to which a patient may be at risk for anticholinergic side effects that can lead to cognitive dysfunction and delirium. The ARS ranks medications for anticholinergic potential on a 3-point scale (0, no or low risk; 3, high anticholinergic potential). The ARS score for a patient is the sum of points for his or her number of medications.

SECONDARY OUTCOMES:
The Fracture Risk Assessment Tool (FRAX) | 1 week after the start of the study
  The FRAX will be used to assess fracture risk in patients. The University of Sheffield launched the FRAX tool in 2008 (Center for Metabolic Bone Diseases, University of Sheffield, UK). It was developed by the FRAX® tool to assess fracture risk in patients. It is based on individual patient models combining fracture risk associated with clinical risk factors and femoral neck bone mineral density (BMD) measurement.
  FRAX® models were developed based on population-based cohort studies conducted in Europe, North America, Asia and Australia.
  FRAX® algorithms provide the 10-year probability of fracture. The result indicates the 10-year probability of having a hip fracture and a major osteoporotic fracture (clinical vertebral, forearm, hip or shoulder fracture).

CONTACTS AND LOCATIONS:
Overall Officials: Bilal UYSAL, assistant prof., Principal Investigator — Balikesir University
Locations (1):
- Balikesir University Health Practice and Research Hospital, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anticholinergic medication use and falls in postmenopausal women: findings from the women's health initiative cohort study